CLINICAL TRIAL: NCT05988827
Title: Effect of Minimizing Light Exposure Intensity of 3D Digital Visualization (NGenuity) on Macular Function After Cataract Surgery in Patients With Early or Intermediate AMD: A Comparative ERG
Brief Title: Effect of Minimizing Light Exposure Intensity on Macular Function After Cataract Surgery in Patients With Early or Intermediate AMD
Acronym: EMERGING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elsan (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023-A00815-40
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Macular Degeneration, Age Related; Cataract
Keywords: Cataract, AMD, light exposure
MeSH Terms: conditions — Macular Degeneration; Cataract

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, 2-arm controlled, parallel, single-masked, single-center study
Who Masked: Participant
Masking Description: Participant is not aware about the light exposure used during the surgery (NGenuity or SOM)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- NGenuity (Experimental): NGenuity allowing a reduced light intensity to 15% during cataract surgery
  Interventions: Device: NGenuity
- SOM (No Intervention): microscope without NGenuity with light intensity of 60%, similar to a Standad Operating Microscope (SOM)

INTERVENTIONS:
Device: NGenuity — Cataract surgery performed under microscope using NGenuity
  Arms: NGenuity

SUMMARY:
Cataract surgery is one of the most frequently performed surgical interventions worldwide. The microscope light-induced retinal toxicity after cataract surgery has been described in several reports even in short procedures; however, this potential toxicity has not been evaluated by objective criteria. Indeed, this retinal phototoxicity would be increased for patients with mild macular diseases such as early stages of AMD (Aged Macular Degeneration) (ie: drusen) which are frequently associated in elderly patients with cataract.

The aim of the study will be to assess the potential functional macular effects by focal and multifocal ERG after cataract surgery with NGenuity by comparison to Standard Operating Microscope (SOM). This study would particularly address eyes at risk for macular toxicity like patients with early or intermediate AMD

DETAILED DESCRIPTION:
Cataract surgery is one of the most frequently performed surgical interventions worldwide. The development of phacoemulsification technology, instrumentation and surgical techniques has improved both the efficacy and safety of procedures, reducing rates of serious postoperative adverse events. The microscope light-induced retinal toxicity after cataract surgery has been described in several reports even in short procedures; however, this potential toxicity has not been evaluated by objective criteria. Indeed, this retinal phototoxicity would be increased for patients with mild macular diseases such as early stages of AMD (Aged Macular Degeneration) (ie: drusen) which are frequently associated in elderly patients with cataract. A systematic literature review of 129 664 individuals estimated the prevalence of early macular degeneration to 8.01% in population aged 45 to 85 years. A three-dimensional (3D) heads-up system (NGenuity®, Alcon, Fort Worth, TX) was recently introduced for both vitreoretinal and cataract surgery, radically improving the quality of surgical visualization. This system allows performing cataract surgery at a lower fraction of light intensity reducing patient's photophobia complaints during surgery and probably preventing potential phototoxic macular injury in cataract surgery. In a recent pilot study, the Ngenuity system was reported to decrease significantly the operative light intensity and to contribute to a faster visual recovery relative to traditional microscopes in series of 35 patients (51 eyes) who underwent cataract surgery. The aim of the study will be to assess the potential functional macular effects by focal and multifocal ERG after cataract surgery with NGenuity by comparison to Standard Operating Microscope (SOM). This study would particularly address eyes at risk for macular toxicity like patients :

* with early AMD: medium-sized drusen (between 63µm and 125µm in diameter) without pigmentary abnormalities
* with intermediate AMD : large drusen (>125 µm) or pigmentary abnormalities in the retina associated with at least medium drusen

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing cataract surgery and presenting signs of early AMD with medium-sized drusen (between 63 µm and 125 µm in diameter) or intermediate AMD with large drusen (>125 µm) or pigmentary abnormalities with at least medium sized drusen in the study eye.
* Patient affiliated to health care system
* Patient with signed informed consent

Exclusion Criteria:

* Children under 18 years old
* AMD defined by geographic atrophy or pigment epithelium detachment, subretinal hemorrhage or visible subretinal new vessel, or subretinal fibrous scars in the study eye
* Non-age-related cataracts
* History of previous ocular surgery, anterior segment (corneal, anterior chamber, sulcus) or posterior segment (uveal, vitreo-retinal) pathology including retinal vascular occlusive disease, retinal detachment or peripheral retinal laser photocoagulation, neovascular AMD, glaucoma in the study eye
* Any current anterior or posterior segment inflammation of any etiology, and/or history of any disease producing an intraocular inflammatory reaction.
* Patient with conditions that increase the risk of zonular rupture during cataract extraction procedure that may affect the postoperative centration or tilt of the IOL
* Patient treated by plaquenil
* Patient already enrolled in the same study for one eye
* Patient already enrolled in clinical trial or with exclusion period in progress
* Patient under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision
* Pregnant or breastfeeding women
* Patient hospitalized without consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-09-14 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-08-09 (Actual)

PRIMARY OUTCOMES:
Assess the change from baseline of the retinal response amplitude in voltage in patients one hour after cataract surgery performed with NGenuity compared to standard light condition with SOM. | 1 hour after cataract surgery
  The change from baseline of the photopic b-wave amplitude (µV) measured one hour after the cataract surgery by fERG.

SECONDARY OUTCOMES:
Assess the change from baseline in both arms of amplitude of the response in voltage in patients one day and one month after cataract surgery | 1 day and 1 month after cataract surgery
  The change from baseline of photopic b-wave amplitude (µV) measured at postoperative day and 1 month after surgery by fERG
Assess the change from baseline in both arms of latency of response in time in patients one hour, one day and one month after cataract surgery | 1 hour, 1 day and 1 month after cataract surgery
  The change from baseline in both arms of fERG implicit time (msec) measured at one hour, one day and one month after cataract surgery
Assess the change from baseline in both arms of total photoreceptors response in the macula one day and one month after cataract surgery | 1 day and 1 month after cataract surgery
  The change from baseline in both arms of Multifocal ERG amplitude (µV) measured at one day and one month after cataract surgery
Assess the change from baseline in both arms of visual acuity one hour, one day and one month after cataract surgery. | 1 hour, 1 day and 1 month after cataract surgery
  The change from baseline in both arms of visual acuity measured on 10 scale one hour, one day and one month after cataract surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Otman Sandali, MD, Principal Investigator — Hopital Prive Guillaume de Varye ELSAN
Locations (1):
- Hopital privé Guillaume de Varye, Saint-Doulchard, France